CLINICAL TRIAL: NCT01111760
Title: Radiation Dose From Computed Tomography Before and After Implementation of a High Pitch Dual Spiral Technique
Acronym: FLASH
Status: Completed | Type: Observational
Sponsor: Michael Gallagher (Other)
Responsible Party: Sponsor-Investigator, Michael Gallagher, Cardiologist, Corewell Health East
Organization: Corewell Health East (Other)
Other Study IDs: HIC 2010-082
Record Dates: First submitted 2010-04-26; First posted 2010-04-28 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Atherosclerosis of Coronary Artery; Cardiovascular Disease; Pulmonary Embolism; Aortic Aneurysm Without Mention of Rupture Nos
Keywords: cardiovascular disease; heart CT scan; CT scan; pulmonary embolisms; aortography
MeSH Terms: conditions — Coronary Artery Disease; Cardiovascular Diseases; Pulmonary Embolism; Aortic Aneurysm

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to compare the radiation exposure of a variety of chest CT examinations performed on the current state of the art CT scanners (64 slice, dual source CT scanner) with the radiation exposure for identical chest CT examinations performed on the Siemens Flash CT scanner (high pitch dual source spiral technique).

DETAILED DESCRIPTION:
Computed tomography has emerged as the "gold standard" for the diagnosis of a broad range of medical diagnoses. For cardiac imaging alone, the installation of CT scanners in US cardiology practices alone has tripled over the past 2 years. Patients who undergo cardiac CTA (computed tomography angiography) may be subjected to relatively high doses of ionizing radiation (ie. 4 times annual background radiation) during the diagnosis and management of coronary artery disease. Current radiation doses for cardiac CT examinations are comparable to the effective doses for patients undergoing nuclear stress tests or cardiac catheterization (ie. approximately 10-15 milliSieverts). In addition, non cardiac CT protocols, such as chest CT examinations for the evaluation of pulmonary arteries, thoracic and abdominal aorta, and lung nodules, are associated with significant radiation exposure. Many patients undergo repeated CT examinations over several years for such pathology. There is a growing public concern regarding the cancer risk associated with such radiation.

Recent major technological advances have been made with the advent of newer generation CT scanners which allow significant radiation dose reduction. One such scanner, the dual source CT, is a new high pitch dual source spiral technique that offers the ability to image a patient's chest with ECG gated imaging protocols within a single second. These technological advances allow significant radiation dose savings, often resulting in effective radiation doses of less than one millisievert (mSv).

ELIGIBILITY:
Inclusion Criteria:

* All patients who undergo chest CT examinations (including cardiac CTA, and non cardiac CT examinations including pulmonary embolism, lung nodule and aortic pathology protocols)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: any patient receiving a coronary CT scan and a chest CT for pulmonary embolisms, pulmonary nodules, aortic pathologies
Sampling Method: Probability Sample
Enrollment: 334 (Actual)
Dates: Start 2010-05; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Comparison of the radiation dose for chest CT examinations using current technology with radiation dose exposure using the newest generation CT scanner. | Time of CT scan
  The primary objective of this study is to compare the estimated radiation dose for chest CT examinations (cardiac and non cardiac) performed using current technology (ie. Retrospective gated CT examinations on the 64 slice and dual source Definition Siemens CT scanners) with the radiation exposure using the newest generation CT scanner (high pitch dual source spiral technique).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gallagher, MD, Principal Investigator — Corewell Health East; Gilbert Raff, MD, Study Director — Corewell Health East
Locations (1):
- William Beaumont Hospital-Royal Oak, Royal Oak, Michigan, United States